CLINICAL TRIAL: NCT02916875
Title: Individual Survivorship Program for Ovarian Cancer Patients Based on PROM's and Shared Decision Making
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Collaborators: Danish Cancer Society (Other); AmbuFlex (Other)
Responsible Party: Sponsor
Other Study IDs: PROMova
Record Dates: First submitted 2016-09-23; First posted 2016-09-28 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Cancer; PROM; Quality of Life
Keywords: Shared decision Making; Follow-up
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In 2015 the Danish healthcare authorities initiated major changes in the follow-up (FU) program for patients with ovarian cancer. The new FU program argues that there is no effect of routine monitoring, and every patient's FU is now individualized. These changes have caused major concern, especially regarding the omission of routine examinations aimed at detection of recurrence, since clinical symptoms of relapse can be diffuse. Clearly, tools and FU plans to support the patients in feeling safe during FU are of vital importance.

Patient-reported outcome measures (PROM) is a tool to improve the focus on patients' needs, symptoms and preferences. It is also a tool to monitor quality of life (QoL), and side effects.

300 patients with ovarian cancer are planned to be enrolled after primary treatment when they enter follow-up program. This is a multi-center study.

All participants fill in a questionnaire at baseline and then every 3 months for two years, and every 6 months the third year. The questionnaire consists of EORTC-QLQ-C30, EORTC-OV28, and questions on symptoms of relapse. At baseline the questionnaire is extended with demographic issues.

The patients will also fill in a brief questionnaire (CollaboRATE) dealing with patient satisfaction and the level of shared decision making experienced.

All participants are followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age.
* Histologically confirmed epithelial ovarian, fallopian tube or serous primary peritoneal cancer.
* Have completed their first line treatment, with complete remission.
* Manage to read and speak Danish.
* Can receive active anti-cancer treatment such as maintenance bevacizumab

Exclusion Criteria:

•Have recurrent disease after first line treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with Ovarian Cancer
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction as measured by combined questionnaires CollaboRATE and Patient Experience. | 3 years.

SECONDARY OUTCOMES:
Quality of life and symptom screening as measured by combined questionnaires EORTC QLQ-C30, EORTC-OV28, and symptom screening questions. | 3 years. Every 3 months for two years and every 6 months the third year.

CONTACTS AND LOCATIONS:
Overall Officials: Anette S. Kargo, MD, Principal Investigator — University of Southern Denmark and Vejle Hospital, Denmark; Karina D. Steffensen, MD, PhD, Study Chair — Vejle Hospital, Denmark
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark

REFERENCES:
- [Derived] Kargo AS, Coulter A, Lindemann K, Jensen PT, Hjollund NH, Mosgaard BJ, Steffensen KD. Use of PROM during follow-up of patients with ovarian cancer: the PROMova study protocol. Int J Gynecol Cancer. 2020 Sep;30(9):1444-1449. doi: 10.1136/ijgc-2020-001528. Epub 2020 Jun 24. PMID 32586892